CLINICAL TRIAL: NCT05179304
Title: Aesthetic Outcomes of Oncoplastic Breast Surgery With a Droplet-Shaped Glandular Flap for Breast Cancer in the Upper Inner Quadrant
Brief Title: Aesthetic Outcomes of Oncoplastic Breast Surgery for Breast Cancer in the Upper Inner Quadrant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shicheng Su, Director of Shuhua Breast Cancer Research Center of Sun Yat-Sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-124-001
Record Dates: First submitted 2021-12-12; First posted 2022-01-05 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Oncoplastic Breast Surgery; Breast Cancer; Aesthetic Outcomes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncoplastic technique with a droplet-shaped glandular flap (Experimental)
  Interventions: Procedure: Oncoplastic technique with a droplet-shaped glandular flap

INTERVENTIONS:
Procedure: Oncoplastic technique with a droplet-shaped glandular flap — A droplet-shaped glandular flap (DSG) is in a shape of a water drop, with the pedicle at the top of the defect and the base underlying nipple-areolar complex (NAC). It runs from the outer upper quadrant to the center along a line parallel to the radial line. We harvest a DSG flap by dissociating the supplement mammary gland from the lateral of the defect after resection, developing deep to the pectoralis fascia, from the cusp at the defect and the round pore underlying nipple-areolar complex (NAC). The DSG flap was rotated inwards around the cusp, reaching the top of the defect. This tailored redistribution allowed the defects to be "plugged" with the lateral glandular flaps.

SUMMARY:
Oncoplastic breast surgery, combining oncological resection with plastic surgical techniques, has emerged as an important surgical strategy to optimize conventional breast-conserving surgery. The upper inner quadrant is one of the most difficult and challenging tumor locations for surgeons to perform oncoplastic breast surgery. There is a pressing need to develop a simple and effective oncoplastic surgical technique to cope with the unfavorable anatomy and location of tumors in the UIQ. Here, we present a new oncoplastic volume displacement technique for UIQ using the DSG flap. This trial was design to estimate the aesthetic outcomes of an oncoplastic technique using a droplet-shaped glandular flap for breast cancer in the upper inner quadrant.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent.
* Female aged between 18 and 70 years.
* Pathologically diagnosed operable breast cancer.
* WHO Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Cancer located in the upper inner quadrant; Single tumor or multiple tumors in the same quadrant.
* The important organ functions meet the following criteria:
* WBC >=3.0 x 10^9/L; Neutrophilic granulocytes >=1.5×10^9/L; Platelet >=100 x 10^9/L; Hb >=9 g/dL;
* Total bilirubin no more than 1.5 times the normal upper limit (ULN); AST and ALT no more than 1.5 times ULN; AKP no more than 2.5 times ULN;
* Serum creatinine no more than 1.5 times ULN or Clearance rate of creatinine >= 60ml/min;
* Thyroid stimulating hormone (TSH) <= ULN (T3, T4 levels need to be detected simultaneously if abnormalities, the patient can be included if T3, T4 levels is normal);
* LVEF basement >= 50%.
* Adjust to the criteria of breast conserving surgery.

Exclusion Criteria:

* Multifocal or multicentric disease.
* Tumor localized in the central quadrant or the distance to the nipple < 2 cm；
* Diffused calcifications with fine plemorphic or fine linear or fine-linear branching morphology.
* The ratio of tumor to breast > 20%;
* The diameter of tumor is up to 4 cm;
* Women in the early or intermediate stage of pregnancy;
* Prior history of breast radiation;
* Any severe comorbidities, inability to give informed consent or unavailability for follow-up.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
aesthetic outcomes | half a year to one year
  ABNSW system. The total score was 15 points, outcomes were good when it was 11-14, fair when it was 6-10, and poor when it was 0-5.

SECONDARY OUTCOMES:
Patients' quality of life | half a year to one year
  EORTC QLQ-C30 questionnaire
Local recurrence | half a year to one year
  Local recurrence defined as histologic evidence of ductal carcinoma in situ or invasive breast cancer in the ipsilateral breast or chest wall.
Patients complications after surgery | half a year to one year
  The occurence of scarring, radiation fibrosis, seroma, fat necrosis and infection

CONTACTS AND LOCATIONS:
Locations (1):
- Shicheng Su, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No